CLINICAL TRIAL: NCT00000880
Title: Phase II Study of Cyclosporin (Neoral) in Immune Activation and HIV Expression in Early HIV Disease
Brief Title: A Study to Test the Effect of Cyclosporine on the Immune System of Patients With Early HIV Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 334; 11306 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: T-Lymphocytes; Lymphocyte Transformation; HIV-1; Drug Therapy, Combination; Immunosuppressive Agents; Apoptosis; Cyclosporine; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections | interventions — Cyclosporine

INTERVENTIONS:
Drug: Cyclosporine

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of low doses of cyclosporine (CsA) in patients with early HIV infection and to evaluate its effect on the immune system.

Activation of T cells (cells of the immune system) leads to HIV replication. Inhibition of immune activation is therefore a potentially important area of therapy for patients with early HIV infection. CsA is capable of decreasing T cell activation, which in turn may decrease HIV replication.

DETAILED DESCRIPTION:
There is increasing data on the potential for inhibition of immune activation as primary therapy for HIV infection. The rationale of CsA therapy is to decrease T cell activation in patients with early HIV infection. Activation of T cells leads to translation and transcription of provirus, release of viral progeny, and ultimately cell death. T cell activation also leads to increased cell death via apoptosis. CsA is capable of inhibiting both these events and thus may lead to decreased CD4 cell turnover.

This study has 2 arms of 15 patients each. Patients in Arm I receive placebo. Patients in Arm II receive CsA. Each arm is further divided into 2 strata. Stratum 1 patients are not allowed to receive antiretroviral therapy. Stratum 2 patients must receive 1 of the following 4 stable nucleoside analogue combinations:

1. Zidovudine (ZDV) plus lamivudine (3TC)
2. ZDV plus didanosine (ddI)
3. Stavudine (d4T) plus 3TC
4. d4T plus ddI.

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this study if you:

* Are HIV-positive.
* Have a CD4 count greater than or equal to 500/mm3.
* Have a plasma HIV RNA level greater than 600 copies/ml.
* Are over 18 years of age.
* Agree to practice abstinence or use barrier methods of birth control during the study.

Exclusion Criteria

You will not be eligible for this study if you:

* Have a history of an AIDS-defining illness, autoimmune disease, or hypertension.
* Have renal disease.
* Have any active infection other than HIV.
* Have used certain antiretroviral medications.
* Are pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Study Completion 2000-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: L Calabrese, Study Chair; M Lederman, Study Chair
Locations (12):
- United States (12):
  - San Francisco Gen Hosp, San Francisco, California
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Northwestern Univ Med School, Chicago, Illinois
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Harvard (Massachusetts Gen Hosp), Boston, Massachusetts
  - Beth Israel Med Ctr, New York, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Case Western Reserve Univ, Cleveland, Ohio
  - Univ of Texas Med Branch, Galveston, Texas
  - Univ of Washington, Seattle, Washington

REFERENCES:
- [Background] Calabrese LH, Lederman MM, Spritzler J, Coombs RW, Fox L, Schock B, Yen-Lieberman B, Johnson R, Mildvan D, Parekh N; AIDS Clinical Trials Group 334 Investigators. Placebo-controlled trial of cyclosporin-A in HIV-1 disease: implications for solid organ transplantation. J Acquir Immune Defic Syndr. 2002 Apr 1;29(4):356-62. doi: 10.1097/00126334-200204010-00005. PMID 11917239